CLINICAL TRIAL: NCT00876005
Title: Perioperative Supplemental Oxygen and the Risk of Surgical Site Infection
Brief Title: Supplemental Oxygen and the Risk of Surgical Site Infection
Acronym: PORSSI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Santa Clara Valley Health & Hospital System (Other)
Responsible Party: Neena Duggal, MD, Santa Clara Valley Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 5/11/07-04
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-05

CONDITIONS: Surgical Site Infection
Keywords: Wound infection
MeSH Terms: conditions — Surgical Wound Infection; Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 80% oxygen during cesarean section
  Interventions: Other: Oxygen by mask
- 2 (Active Comparator): 30% oxygen during cesarean section
  Interventions: Other: Oxygen by mask

INTERVENTIONS:
Other: Oxygen by mask — Postoperatively, an aerosol face mask is used to deliver oxygen at 80%
  Other Names: Face mask delivery of supplemental oxygen at 80%
  Arms: 1
Other: Oxygen by mask — Postoperatively, an aerosol face mask is used to deliver oxygen at 30%
  Other Names: face mask delivery of supplemental oxygen at 30%
  Arms: 2

SUMMARY:
This is a study to see whether increasing the oxygen concentration during and after a cesarean section decreases the infection rate.

DETAILED DESCRIPTION:
This is a double-blinded prospective randomized,controlled trial to evaluate whether using a higher concentration of oxygen during and after surgery helps to decrease the wound infection rate in patients undergoing cesarean sections.

ELIGIBILITY:
Inclusion Criteria:

* mentally competent patients undergoing cesarean section under spinal or epidural anesthesia

Exclusion Criteria:

* fever/chorioamnionitis; GBS positive on antibiotics; immunocompromised / HIV patients; on antibiotics for any reason; general anesthesia; age less than 18 years custody patients stat cesarean section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1202 (Estimated)
Dates: Start 2006-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neena Duggal, MD, Principal Investigator — Santa Clara Valley Medical Center
Locations (1):
- Santa clara Valley Medical Center, San Jose, California, United States

REFERENCES:
- [Derived] Duggal N, Poddatorri V, Noroozkhani S, Siddik-Ahmad RI, Caughey AB. Perioperative oxygen supplementation and surgical site infection after cesarean delivery: a randomized trial. Obstet Gynecol. 2013 Jul;122(1):79-84. doi: 10.1097/AOG.0b013e318297ec6c. PMID 23743467